CLINICAL TRIAL: NCT04915508
Title: Extremely Hypofractionated Intensity Modulated Stereotactic Body Radiotherapy for Adjuvant or Salvage Treatment for Rising PSA After Radical Prostatectomy (EXCALIBUR)
Brief Title: Extremely Hypofractionated Intensity Modulated Stereotactic Body Radiotherapy for the Treatment of Prostate Cancer With Rising PSA After Radical Prostatectomy
Acronym: EXCALIBUR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-000263; NCI-2021-05447 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Prostate Adenocarcinoma; Stage IIIB Prostate Cancer American Joint Committee on Cancer (AJCC) v8; Stage IIIC Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8; Stage IVA Prostate Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Steroids; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment (SBRT, hormone therapy) (Experimental): Patients undergo SBRT every other day or on consecutive days for up to 14 days. Patients may receive hormonal therapy at the discretion of the treating physician.
  Interventions: Drug: Hormone Therapy; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Drug: Hormone Therapy — Receive hormonal therapy
  Other Names: Chemotherapy-Hormones/Steroids; Endocrine Therapy; Hormonal Therapy; hormone treatment
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase II trial investigates the effect of extremely hypofractionated intensity modulated stereotactic body radiotherapy in treating patients with prostate cancer that has rising prostate specific antigen (PSA) after radical prostatectomy. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the two-year change in patient-reported gastrointestinal (GI) symptoms based on the Expanded Prostate Cancer Index (EPIC) instrument following stereotactic body radiotherapy (SBRT) to the prostate bed and/or pelvic lymph nodes, with a comparison to historical control data for more prolonged radiation regimens.

II. To determine the two-year change in patient-reported urinary (GU) symptoms based on the EPIC instrument following stereotactic body radiotherapy (SBRT) to the prostate bed and/or pelvic lymph nodes, with a comparison to historical control data for more prolonged radiation regimens.

SECONDARY OBJECTIVES:

I. To quantify patient-reported GI symptoms using the EPIC instrument at 3 months, 6 months, 1 and 5 years.

II. To quantify patient-reported GU symptoms using the EPIC instrument at 3 months, 6 months, 1 and 5 years.

III. To quantify rates and severity of acute physician scored adverse events using the Common Terminology Criteria for Adverse Events (CTCAE version [v.] 5.0) scale.

IV. To quantify the five-year cumulative incidence of physician scored adverse events the CTCAE v4.03 scale.

V. To quantify five-year progression-free survival. VI. To quantify 5-year cumulative incidence of biochemical recurrence. VII. To quantify 5-year distant metastasis-free survival.

EXPLORATORY OBJECTIVES:

I. To compare all primary and secondary endpoints between patients treated with an magnetic resonance imaging (MRI)-guided versus a computed tomography (CT)-guided linear accelerator.

II. To compare primary and secondary endpoints between patients treated with short course (=< 6 months) or long-term >= 12 months) antiandrogen therapy (ADT).

OUTLINE:

Patients undergo SBRT every other day or on consecutive days for up to 14 days. Patients may receive hormonal therapy at the discretion of the treating physician.

After completion of study treatment, patients are followed up every 3 months for the first year, and then every 6 months for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* History of histologically confirmed, clinical localized adenocarcinoma of the prostate treated with radical prostatectomy with definitive intent
* Presence of any ONE of the following:

  * Adverse pathologic features at the time of prostatectomy (positive surgical margin, pathologic T-stage 3-4 disease, pathologic Gleason score 8-10 disease, OR presence of tertiary Gleason grade 5 disease)
  * Documentation of rising prostate-specific antigen on at least two consecutive draws, with the magnitude of prostate-specific antigen exceeding 0.03 ng/mL
  * Intermediate- or high-risk Decipher genomic classifier score
  * Identification of prostate cancer in >= 1 lymph node at the time of prostatectomy (pN+ disease)
* CT scan and MRI of the pelvis within 120 days prior to enrollment [note: (a) if patient has medical contraindication to MRI, an exemption will be granted and enrollment can proceed; (b) for patients with PSA < 1.0 ng/mL, the treatment planning CT can substitute for a diagnostic CT scan; (c) a low-field, radiation planning MRI can replace the diagnostic MRI if the patient refuses or cannot obtain a high-field MRI]
* Bone scan OR advanced nuclear imaging study within 120 days prior to enrollment for patients with PSA > 1.0 ng/mL
* Age >= 18
* Karnofsky performance status (KPS) >= 70 and/or Eastern Cooperative Oncology Group (ECOG) =< 2
* Ability to understand, and willingness to sign, the written informed consent

Exclusion Criteria:

* Patients with any evidence of distant metastases. Note, evidence of lymphadenopathy below the level of the renal arteries can be deemed loco regional per the discretion of the investigator
* Patients with neuroendocrine or small cell carcinoma of the prostate
* Prior pelvic radiotherapy
* History of Crohn's disease, ulcerative colitis, or ataxia telangiectasia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2021-06-23 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2027-08-01 (Estimated)

PRIMARY OUTCOMES:
Change of Expanded Prostate Cancer Index (EPIC) score for the gastrointestinal domain | Baseline up to 2 years
  EPIC assessed the disease-specific aspects of prostate cancer and its therapies within the gastrointestinal summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
Change of Expanded Prostate Cancer Index (EPIC) score for the genitourinary domain | Baseline up to 2 years
  EPIC assessed the disease-specific aspects of prostate cancer and its therapies within the genitourinary summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.

SECONDARY OUTCOMES:
Patient-reported gastrointestinal (GI) symptoms | At 3 months, 6 months, 1year, and 5 years
  EPIC assessed the disease-specific aspects of prostate cancer and its therapies within the gastrointestinal summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
Patient-reported genitourinary (GU) symptoms | At 3 months, 6 months, 1year, and 5 years
  EPIC assessed the disease-specific aspects of prostate cancer and its therapies within the genitourinary summary domain. Response options for each EPIC item formed a Likert scale, and multi-item scale scores were transformed linearly to a 0-100 scale, with higher scores representing better Health-Related QoL.
Incidence of acute physician scored adverse events | Up to 5 years
  Will be assessed by using the Common Terminology Criteria for Adverse Events version 4.0.
Cumulative incidence of physician scored adverse events | Up to 5 years
  Will be assessed by using the Common Terminology Criteria for Adverse Events version 4.0.
Progression-free survival | Up to 5 years
Cumulative incidence of biochemical recurrence | Up to 5 years
Distant metastasis-free survival | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Amar Kishan, Principal Investigator — UCLA / Jonsson Comprehensive Cancer Center
Locations (1):
- UCLA / Jonsson Comprehensive Cancer Center, Los Angeles, California, United States